CLINICAL TRIAL: NCT04486105
Title: Investigation of Sucrose-induced Metabolic Adaptation and Biomarkers of Chronic Sucrose Intake in Humans Using a Multi-omic Approach
Brief Title: Chronic Sucrose Intake, Markers of Health and Biomarker Identification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, John Lodge, Associate Professor, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 15738
Record Dates: First submitted 2020-07-15; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Dietary Exposure; Metabolic Disturbance
MeSH Terms: interventions — Sucrose

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (Placebo Comparator): vehicle only for one week
  Interventions: Dietary Supplement: sucrose
- 40g sucrose ingestion (Experimental): 40g sucrose treatment on top of habitual diet for one week
  Interventions: Dietary Supplement: sucrose
- 80g sucrose ingestion (Experimental): 80g sucrose treatment on top of habitual diet for one week
  Interventions: Dietary Supplement: sucrose
- 120g sucrose ingestion (Experimental): 120g sucrose treatment on top of habitual diet for one week
  Interventions: Dietary Supplement: sucrose

INTERVENTIONS:
Dietary Supplement: sucrose — pure sucrose in water in addition to habitual diet

SUMMARY:
With free sugar intake proving to be of a concern within the general public, discovery and validation of a new biomarker will allow for more consistent measurement of sucrose intake. Furthermore, using a multi-omic approach the investigators will identify metabolic perturbations to the metabolome and proteome.

DETAILED DESCRIPTION:
Excessive free sugar intake is of concern within the general public, as intakes have been associated with weight gain and cardiovascular disease. Average intakes are over double that of the 5% of total energy intake that is recommended by the Science Advisory Committee on Nutrition, but intakes are calculated from observational measures that lack sensitivity and discovery and validation of a new biomarker from biological fluids may allow for more specific measurement and a better understanding of intake:disease relationships. Furthermore, understanding the biochemistry of sucrose intake will allow the identification of damage occurrence and alternative metabolic pathways, as well as novel protein damage that occur with chronic sucrose exposure.

This study aims to identify a biomarker of chronic sucrose consumption using metabolite profiling technology. The study will be composed of a randomised controlled intervention trial, in which participants will be required to consume an amount of sucrose (0-120g/d) every day for 7 days and provide biofluid samples (urine and blood) before the initiation, during and following the intervention; that will undergo metabolic analysis. Furthermore, participants will have their anthropometrics and dietary intake monitored throughout the study. The biomarker will also be validated against the dietary information and correlated with indices of health and sucrose-induced damage. The investigators will also monitor the feasibility and acceptability of chronic sucrose intake during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-64, healthy diagnosis

Exclusion Criteria:

* gastrointestinal issues, doesn't consume sugar

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | change in blood pressure following one week intervention
  Measurement of systolic and diastolic blood pressure
Metabolome | change in the urinary metabolome following one week intervention
  Metabolite profiling of urine samples, obtaining a profile of approximately 5000 metabolite intensities in urine
Body composition | change in body mass index following one week intervention
  measurement of body mass index
Body composition | change in percentage body fat following one week intervention
  measurement of percentage body fat

SECONDARY OUTCOMES:
food diary analysis | change in dietary intake following the week intervention
  measurement of energy, macro and micronutrient intakes from 3-day food diaries

CONTACTS AND LOCATIONS:
Overall Officials: John Lodge, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumberland Building, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No